CLINICAL TRIAL: NCT05412979
Title: A Multicenter, Randomized, Double-Blind, Crossover, Phase 2 Study Evaluating the Safety and Efficacy of Hormone Replacement Therapy With ST-1891 Compared to Levothyroxine in Patients With Primary Hypothyroidism
Brief Title: A Study Evaluating the Safety and Efficacy of Hormone Replacement Therapy With ST-1891 Compared to Levothyroxine in Patients With Primary Hypothyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sention Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-1891-201
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ST-1891 (Experimental)
  Interventions: Drug: ST-1891
- Levothyroxine (Active Comparator)
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: ST-1891 — ST-1891
  Arms: ST-1891
Drug: Levothyroxine — Levothyroxine
  Arms: Levothyroxine

SUMMARY:
ST-1891-201 is a multicenter, randomized, double-blind, partial crossover, Phase 2 study evaluating the safety and efficacy of hormone replacement therapy with ST-1891 compared to levothyroxine in patients with primary hypothyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary hypothyroidism
* On continuous thyroid replacement therapy with levothyroxine for at least 12 months immediately prior to Screening
* On a stable daily dose of levothyroxine for the 3 months prior to Screening
* Willing to give written informed consent for the Study

Exclusion Criteria:

* Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation or excretion of ST-1891 or levothyroxine
* Female patients who are pregnant or are breastfeeding starting 30 days prior to Screening
* Anticipated initiation or change in concomitant medications
* Concomitant use of prohibited medications
* Currently participating in another clinical study or have received active treatment with an investigational drug within 30 days or 5 half-lives of the investigational drug of Screening, whichever is longer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Levothyroxine-to-ST-1891 dosing conversion factor | Week 52

SECONDARY OUTCOMES:
Percent of patients with a thyroid-stimulating hormone (TSH) level within the standard reference range | Week 52
Time to TSH normalization | Week 52

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Sention Investigational Site, Greenbrae, California
  - Sention Investigational Site, Newhall, California
  - Sention Investigational Site, Denver, Colorado
  - Sention Investigational Site, Fort Lauderdale, Florida
  - Sention Investigational Site, Jacksonville, Florida
  - Sention Investigational Site, New Port Richey, Florida
  - Sention Investigational Site, Palm Harbor, Florida
  - Sention Investigational Site, Atlanta, Georgia
  - Sention Investigational Site, Lawrenceville, Georgia
  - Sention Investigational Site, Roswell, Georgia
  - Sention Investigational Site, Evergreen Park, Illinois
  - Sention Investigational Site, Newburgh, Indiana
  - Sention Investigational Site, South Bend, Indiana
  - Sention Investigational Site, Ankeny, Iowa
  - Sention Investigational Site, Louisville, Kentucky
  - Sention Investigational Site, Dearborn, Michigan
  - Sention Investigational Site, Chesterfield, Missouri
  - Sention Investigational Site, Jefferson City, Missouri
  - Sention Investigational Site, Staten Island, New York
  - Sention Investigational Site, Cary, North Carolina
  - Sention Investigational Site, Greenville, North Carolina
  - Sention Investigational Site, Hickory, North Carolina
  - Sention Investigational Site, Morehead City, North Carolina
  - Sention Investigational Site, Raleigh, North Carolina
  - Sention Investigational Site, Rocky Mount, North Carolina
  - Sention Investigational Site, Salisbury, North Carolina
  - Sention Investigational Site, Wilmington, North Carolina
  - Sention Investigational Site, Mt. Pleasant, South Carolina
  - Sention Investigational Site, Bristol, Tennessee
  - Sention Investigational Site, Chattanooga, Tennessee
  - Sention Investigational Site, Memphis, Tennessee
  - Sention Investigational Site, Austin, Texas
  - Sention Investigational Site, Benbrook, Texas
  - Sention Investigational Site, Live Oak, Texas
  - Sention Investigational Site, Round Rock, Texas
  - Sention Investigational Site, Webster, Texas
  - Sention Investigational Site, Virginia Beach, Virginia
  - Sention Investigational Site, Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided